CLINICAL TRIAL: NCT05604859
Title: Evaluate the Efficacy and Safety of Various Treatment Schemes for Severe Fever With Thrombocytopenia Syndrome：a Prospective, Multicenter, Non-randomized Controlled Intervention Study
Brief Title: Evaluate the Efficacy and Safety of Various Treatment Schemes for Severe Fever With Thrombocytopenia Syndrome(SFTS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNBRELLA STUDY
Record Dates: First submitted 2022-10-31; First posted 2022-11-03 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Severe Fever With Thrombocytopenia Syndrome
Keywords: interleukin-6; D-D dimer; efficacy; safety; severe SFTS
MeSH Terms: conditions — Severe Fever with Thrombocytopenia Syndrome | interventions — Methylprednisolone; Immunoglobulins, Intravenous; tocilizumab; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-intervening group (Active Comparator): conventional treatment，including symptomatic and supportive treatment, antiviral treatment etc.
  Interventions: Other: conventional treatment
- intervention group (Experimental): Part A group: Patients received methylprednisolone 1-2mg/kg/d（or other glucocorticoid equivalent to methylprednisolone 1-2mg/kg/d) + IVIG 0.2g-0.4g/kg/d for a total of 3-5 days. If the disease progressed after treatment, the patients were given the dose of rescue therapy (methylprednisolone > 2mg/kg/d or other glucocorticoid equivalent to methylprednisolone > 2mg/kg/d + IVIG 0.4g/kg/d) for another 3-5 days.
  Part B group: Patients received tocilizumab 4mg/kg once.
  Part C group: Patients received low molecular weight heparin 100U/kg, qd or q12h IH for 4-7 days.
  All patients received conventional treatment. All patients were followed up from the end of treatment to day 28 after completion of treatment.
  Interventions: Drug: Methylprednisolone; Drug: intravenous immunoglobulin; Drug: Tocilizumab; Drug: Low molecular weight heparin; Other: conventional treatment

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone:1-2mg/kg/d(or other glucocorticoid equivalent to methylprednisolone 1-2mg/kg/d),ivgtt,3-5 days.If disease progression occurs after completion of treatment, the dose of salvage therapy (methylprednisolone > 2mg/kg/d or other glucocorticoid equivalent to methylprednisolone > 2mg/kg/d) was continued for another 3-5 days.
  Arms: intervention group
Drug: intravenous immunoglobulin — intravenous immunoglobulin:0.2g-0.4g/kg/d,ivgtt, 3-5 days.If disease progression occurs after completion of treatment, the dose of salvage therapy (IVIG 0.4g/kg/d) was continued for another 3-5 days.
  Arms: intervention group
Drug: Tocilizumab — Tocilizumab:4mg/kg, once
  Arms: intervention group
Drug: Low molecular weight heparin — Low molecular weight heparin:100U/kg, qd or q 12h,IH,4-7 days
  Arms: intervention group
Other: conventional treatment — conventional treatment，including symptomatic and supportive treatment, antiviral treatment etc.

SUMMARY:
This is a prospective, multicenter, non-randomized, controlled intervention clinical study.Patients with severe fever with thrombocytopenia syndrome who have been clinically diagnosed and met the study inclusion criteria will be included in the study for analysis.

All patients with SFTS will be assigned to different groups according to the ratio of 1:3, including the non-intervention group (conventional treatment group) and the related drug intervention group.

Non-intervention group:patients received conventional treatment during hospitalization.

Intervention group:

Part A group: Patients received methylprednisolone 1-2mg/kg/d（or other glucocorticoid equivalent to methylprednisolone 1-2mg/kg/d) + intravenous immunoglobulin (IVIG) 0.2g-0.4g/kg/d for a total of 3-5 days. If the disease progressed after treatment, the patients was given the dose of rescue therapy (methylprednisolone > 2mg/kg/d or other glucocorticoid equivalent to methylprednisolone > 2mg/kg/d + IVIG 0.4g/kg/d) for another 3-5 days.

Part B group: Patients received tocilizumab 4mg/kg once.

Part C group: Patients received low molecular weight heparin 100U/kg, qd or q12h IH for 4-7 days. If the platelet count is less than 30 × 10^9/L, the low molecular weight heparin should be discontinued.

All patients received conventional treatment. All patients were followed up from the end of treatment to day 28 after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years. 2. SFTS Patients met the following diagnostic criteria:SFTS-virus (SFTSV) positive in peripheral blood detected by RT-PCR or Next Generation Sequencing (NGS) .

3. The intervention group shall meet the following conditions:

1. Part A: Treatment can be initiated if the patient has two of the following conditions: (1) Persistent high fever for 7 days or more; (2) Platelets less than 50×10^9/L; (3) Multiple organ function impairment (MODS) including brain, heart, liver, kidney and blood coagulation; (4) Failure of more than 1 organ, such as brain, heart, liver, kidney and coagulation.
2. Part B: Serum cytokine IL-6 quantification >2 times the upper limit of normal (ULN).
3. Part C: Plasma D-D dimer ≥ 4×ULN. 4. Sign written informed consent and cooperate with follow-up.

Exclusion Criteria:

1. Patients with neoplastic diseases.
2. Patients with severe chronic diseases, such as chronic kidney disease stage 3-5, chronic heart failure, decompensated cirrhosis, chronic diseases of the central nervous system, hematologic neoplastic diseases, uncontrolled solid tumors, etc.
3. Patients who are or may be pregnant.
4. Patients with a history of hypersensitivity reaction to the trial drug and its components.
5. Patients with conditions that the investigator judged to affect short-term survival.

Additional exclusion criteria for Part B:

Patients with platelet < 50×10^9/L

Additional exclusion criteria for Part C:

1. Received vasopressor therapy for more than 36 hours before enrollment;
2. Indications for anticoagulant therapy (such as ACS, acute VTE, mechanical valve, etc.);
3. Significant bleeding risk as evidenced by one of the following conditions:

   Clinical: Surgery that requires general or spinal anesthesia within 24 hours prior to enrollment, or may require such surgery within the next 24 hours; Evidence of active bleeding; A history of severe head trauma requiring hospitalization; History of intracranial surgery or stroke or any cerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass within 3 months prior to the study; History of congenital hemorrhage; Gastrointestinal bleeding occurred within 6 weeks before the study unless corrective surgery was performed; Trauma that is thought to increase the risk of bleeding; The presence of an epidural catheter; Laboratory: INR > 2.0, or thrombelastogram results suggest significant hyperfibrinolysis.
4. Present with other forms of shock that are clinically apparent, including cardiogenic, obstructive (massive pulmonary embolism, cardiac tamponade, tension pneumothorax), hemorrhagic, neurogenic, or anaphylactic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
28-day survival rate | From enrollment to 28 day
  28-day survival rate was defined as the proportion of patients who were still alive 28 days after enrollment.

SECONDARY OUTCOMES:
Incidence of complications | From enrollment to 28 day
  The complications include Respiratory system, gastrointestinal system, blood system, nervous system, liver and kidney, lymphatic system, multiple organ dysfunction syndrome may be related to Severe Fever With Thrombocytopenia Syndrome.Incidence of complications was defined as the proportion of complications occur after enrollment.
Incidence of AEs | From enrollment to 28 day
  Incidence of adverse events associated with trial drug treatment: blood glucose, electrolyte disturbances, osteoporosis, Cushing's syndrome, double infection, active bleeding, etc.

OTHER OUTCOMES:
Biomarkers associated with efficacy | From enrollment to 12 month
  Blood, bone marrow, lymph node, urine and stool samples were collected to explore biomarkers associated with predicting the efficacy of methylprednisolone combined with IVIG, tocilizumab and low molecular weight heparin in the treatment of severe fever with thrombocytopenia syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Qin, MD., PhD, Study Chair — Department of Infectious Disease, Tongji Hospital, Tongji Medical College, HUST
Locations (10):
- China (10):
  - Guangshui First Peoples Hospital, Guangshui, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - Luotian County Peoples Hospital, Huanggang, Hubei
  - Macheng Peoples Hospital, Macheng, Hubei
  - Qianjiang Central Hospital, Qianjiang, Hubei
  - Suizhou Central Hospital, Suizhou, Hubei
  - Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - Yichang Third Peoples Hospital, Yichang, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu